CLINICAL TRIAL: NCT04962477
Title: Understanding Host-pathogen Interaction in the Respiratory Mucosa During Pregnancy
Status: Completed | Type: Observational
Sponsor: Washington University School of Medicine (Other)
Responsible Party: Principal Investigator, Arvind Palanisamy, Associate Professor of Anesthesiology, Obstetrics and Gynecology, Washington University School of Medicine
Other Study IDs: 202107016
Record Dates: First submitted 2021-07-02; First posted 2021-07-15 (Actual); Last update posted 2025-12-19 (Actual); Status verified 2025-12

CONDITIONS: Pregnancy Related; Innate Inflammatory Response
MeSH Terms: conditions — Inflammation

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Nasal brush samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Pregnant
  Interventions: Other: Nasal brush sampling
- Non-pregnant
  Interventions: Other: Nasal brush sampling

INTERVENTIONS:
Other: Nasal brush sampling — Nasal brush samples will be collected from the inferior turbinate using standardized techniques after local anesthetic application. After clearing the mucus from the nasal cavity by asking the patient to blow their nostrils twice followed by local anesthetic spray application, nasal brush samples will be collected from the inferior turbinate of each nostril with dedicated soft cytology brushes and pooled together for molecular biological experiments. Simultaneously, 10 mL of peripheral blood will be collected for immunophenotyping.

SUMMARY:
The clinical presentation of the ongoing coronavirus disease-19 (COVID-19) pandemic in pregnant women is unique with more asymptomatic infection, higher morbidity when symptomatic, yet without a difference in mortality rate. This is strikingly different from the high mortality observed during the past influenza A pandemics. Though both influenza A virus (IAV) and SARS-CoV-2 are single-stranded RNA viruses, the exquisite vulnerability of pregnant women to influenza A but not COVID-19 remains a mystery. Our objective, therefore, is to determine the mechanisms that predispose pregnant women to severe influenza A but confer protection against SARS-CoV-2 infection by examining the viral entry factors and innate immune response mechanisms in the nasal epithelium of pregnant vs. non-pregnant age-matched women.

ELIGIBILITY:
Inclusion Criteria:

* Healthy, uncomplicated pregnant subjects in the third trimester ((≥ 28 ≤ 41 weeks' gestation)
* Healthy non-pregnant adult female volunteers between the ages of 18 - 45 years.
* Between 18-45 years old
* Able to provide consent

Exclusion Criteria:

* Patients in labor
* Critically ill patients needing intubation and mechanical ventilation
* Patients with fever or influenza-like illness
* H/o epistaxis or rhinosinusitis
* Nasal polyposis and deviated nasal septum
* Preeclampsia and chronic hypertension
* Use of anti-hypertensives
* Ongoing seasonal allergy
* H/o asthma
* Recent recovery from SARS-CoV-2 or influenza A infection (≤ 4 weeks)
* Recent receipt of either COVID-19 or influenza A vaccine (≤ 4 weeks)
* Use of immunosuppressive medications
* Use of inhaled corticosteroids
* Use of hormonal contraceptives in non-pregnant population
* Allergy to local anesthetic

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Only females are eligible for the study.
Study Population: Pregnant cohort: pregnant women in their third trimester admitted to the hospital for any elective procedure (cesarean delivery, labor induction etc.,)
  Non-pregnant cohort: age-matched female volunteers
Sampling Method: Non-Probability Sample
Enrollment: 48 (Actual)
Dates: Start 2022-03-02 (Actual); Primary Completion 2023-09-27 (Actual); Study Completion 2023-09-27 (Actual)

PRIMARY OUTCOMES:
Expression of viral entry factors | Dec 2021

SECONDARY OUTCOMES:
Expression of genes involved in innate immune response and host-pathogen interaction | Dec 2021

CONTACTS AND LOCATIONS:
Overall Officials: Arvind Palanisamy, MD, Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University in St. Louis, St Louis, Missouri, United States

IPD SHARING:
Plan to Share IPD: No